CLINICAL TRIAL: NCT02384486
Title: Evaluating the Efficacy of a Proposed Training Programme to Reduce Stress in Mothers of Children With Autism Spectrum Disorder (ASD) in Saudi Arabia: A Pilot Study
Brief Title: Efficacy of Training Programme to Reduce Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: OVS12022015 SA SoM PAPsych PhD
Record Dates: First submitted 2015-03-04; First posted 2015-03-10 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Autism Spectrum Disorder (ASD)
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- intervention group (Experimental): intervention group will receive the "Training to Reduce Stress in Mothers of Children with (ASD)"
  Interventions: Behavioral: Training to Reduce Stress in Mothers of Children with (ASD)
- control group (Other): control group will receive nothing but for ethical purposes will receive the same intervention after the end of the trial for the intervention group
  Interventions: Other: Nothing (treatment as usual)

INTERVENTIONS:
Behavioral: Training to Reduce Stress in Mothers of Children with (ASD) — The main objective of the proposed study is to examine the effect of implementing the proposed intervention on stress in mothers of children with ASD in SA
  Arms: intervention group
Other: Nothing (treatment as usual) — Mothers in the control group will continue to receive treatment as usual during the trial
  Arms: control group

SUMMARY:
This study aims to reduce stress in mothers of children with autism in Saudi Arabia. The researcher has designed a training programme for mothers whose children are young and just in their early stage at the autism organisations they are attending. The programme will include stress reduction tips, behavioural modification strategies for children with autism, and financial resources available to parents (how they can access government funding). The study will have two parts. Part one involves conducting an experiment by dividing the participants into two groups, one group will receive the training and the other group will wait until the end of the study then they will also receive the same training. Both groups will fill questionnaire at the beginning of the study, then after the first group finishes training, and then again 6 weeks later. Part two of the study will involve interviewing mothers of the first group who attended the training session. They will be interviewed by the researcher asking them about their experience with the training programme and their suggestions for future improvements. Mothers will be given a training manual at the beginning of the training. Training involves attending five sessions, one of which is a face to face session at the autism organisation their children are attending and the other four sessions will be through a Smartphone application called whatsapp which is widely used in Saudi Arabia.

ELIGIBILITY:
Inclusion Criteria:

* Mothers aged 18 years or over
* mothers of ASD children who are in the early intervention stage (first year in the programme) at autism organizations in Saudi Arabia

Exclusion Criteria:

* Mothers whose children with ASD are not in the early intervention stage or did not joint autism organization

  * Mothers who will not be willing to commence to the full duration of the trial
  * Mothers who will not be able to use whatsapp in their smart phones

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2015-04; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Parent Stress Index Short From (PSI-SF) | 10 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Voluntary sector ASD organization no.1, Jeddah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hemdi A, Daley D. The Effectiveness of a Psychoeducation Intervention delivered via WhatsApp for mothers of children with Autism Spectrum Disorder (ASD) in the Kingdom of Saudi Arabia: A randomized controlled trial. Child Care Health Dev. 2017 Nov;43(6):933-941. doi: 10.1111/cch.12520. Epub 2017 Sep 20. PMID 28929582